CLINICAL TRIAL: NCT05227768
Title: A Dose-escalation, Single-center, Randomized, Double-blinded, Placebo-controlled, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profiles of VV116 Administered Orally to Chinese Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Single Ascending Doses of VV116 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VV116-01
Record Dates: First submitted 2021-12-29; First posted 2022-02-07 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects
Keywords: VV116; Phase I; dose-escalation; Tolerability; Pharmacokinetic
MeSH Terms: interventions — GS-621763; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VV116 (Experimental): Subjects will receive VV116 orally for single dose.
  Interventions: Drug: VV116 25mg Group; Drug: VV116 200mg Group; Drug: VV116 400mg Group; Drug: VV116 800mg Group; Drug: VV116 1200mg Group
- Placebo (Experimental): Subjects will receive placebo orally for single dose.
  Interventions: Drug: VV116 25mg Group; Drug: VV116 200mg Group; Drug: VV116 400mg Group; Drug: VV116 800mg Group; Drug: VV116 1200mg Group

INTERVENTIONS:
Drug: VV116 25mg Group — 4 subjects will receive VV116 25mg,orally; 2 subjects will receive placebo,orally.
  Other Names: Placebo
Drug: VV116 200mg Group — 6 subjects will receive VV116 200mg,orally; 2 subjects will receive placebo,orally.
  Other Names: Placebo
Drug: VV116 400mg Group — 6 subjects will receive VV116 400mg,orally; 2 subjects will receive placebo,orally.
  Other Names: Placebo
Drug: VV116 800mg Group — 6 subjects will receive VV116 800mg,orally; 2 subjects will receive placebo,orally.
  Other Names: Placebo
Drug: VV116 1200mg Group — 6 subjects will receive VV116 1200mg,orally; 2 subjects will receive placebo,orally.
  Other Names: Placebo

SUMMARY:
The study consists of 5 dose groups, starting at 25 mg, 6 subjects in 25 mg group, and 8 subjects in each other group (male or female), randomly assigned to study drug or placebo group to evaluate the safety, tolerability and PK characteristics. The subject number of single dose group may increase or decrease depending on the safety and PK data obtained. The dose levels are planned at 25 mg, 200 mg, 400 mg, 800 mg and 1200 mg. Based on observed tolerability and safety data or obtained PK data, adjustments are allowed at all dose levels in the clinical trial.

DETAILED DESCRIPTION:
4 subjects in the 25 mg dose group will receive VV116 tablets and the other 2 subjects will receive placebo. In other dose groups, 6 subjects in each group will receive VV116 tablets and 2 subjects will receive placebo. 25mg,800mg and 1200 mg dose group will be given by sentinel administration (i.e. 1 study drug, 1 placebo). Subjects who receive sentinel administration will be observed for 48 hours and investigator will evaluate the safety parameters (including symptoms, vital signs, physical examination, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 45 years;
2. Body weight no less than 50 kg for male, no less than 45 kg for female; Body Mass Index of 19 to 26kg/m2;
3. Physical examination, vital signs examination, laboratory examination, ECG, B-ultrasound and fundus examination results were normal or abnormal without clinical significant;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form;

Exclusion Criteria:

1. Subjects with hypersensitivity to VV116 or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with central nervous system,cardiovascular system,gastrointestinal, respiratory system,urinary,Hematologic System,metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
4. Blood donation or blood loss ≥ 400 mL within 3 months prior to inclusion, or have a history of blood product use history;
5. Participated in a clinical study involving another investigational drug within 3 month before the screening visit;
6. Taken any prescription drugs, non-prescription drugs, Chinese herbal medicine or health care products within 2 weeks prior to screening;
7. Drug or alcohol addicts within 1 year prior to screening, who drink at least twice a day or more than 14 units per week, or who are addicted to alcohol (1 unit ≈200 mL beer with 5% alcohol content, 25 mL spirits with 40% alcohol content or 85 mL wine with 12% alcohol content) ;
8. Those who smoke more than 10 cigarettes per day and do not agree to avoid using any tobacco products during the trial period;
9. Those who cannot quit smoking or drinking during the trial;
10. Those who are positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
11. Abnormal and clinically significant chest radiographs (anteroposterior);
12. B ultrasound examination showed moderate to severe fatty liver;
13. Pregnant or lactating women or male subjects whose spouse has a child care plan within 3 months;
14. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 7 days after treatment
  Incidence of Treatment-Emergent Adverse Events
Tmax | From time zero up to 48 hours post-dose following oral administration of VV116
  time at which Cmax occurs
Cmax | From time zero up to 48 hours post-dose following oral administration of VV116
  maximum observed plasma concentration
AUC0~t | From time zero up to 48 hours post-dose following oral administration of VV116
  area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | From time zero up to 48 hours post-dose following oral administration of VV116
  area under the plasma concentration-time curve from time zero to infinity

SECONDARY OUTCOMES:
structural of metabolites | From time zero up to 72 hours post-dose following oral administration of VV116
  Structure of main metabolites of VV116 in plasma, feces and urin. The main metabolites may include 116-N1 and M2.
Ae(total excretion of kidney) | From time zero up to 72 hours post-dose following oral administration of VV116
  Ae(total excretion of kidney)
Ae%(proportion of excretion of kidney) | From time zero up to 72 hours post-dose following oral administration of VV116
  Ae%(proportion of excretion of kidney)
CLr(renal clearance rate) | From time zero up to 72 hours post-dose following oral administration of VV116
  CLr(renal clearance rate)
Cumulative excretion and percentage of VV116 and major metabolites in feces. | From time zero up to 72 hours post-dose following oral administration of VV116
  Cumulative excretion and percentage of VV116 and major metabolites in feces.

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No